CLINICAL TRIAL: NCT05051566
Title: A Multiple Dose Study in Healthy Participants to Investigate the Safety, Tolerability, and Pharmacokinetics of LY3502970
Brief Title: A Multiple Dose Study of LY3502970 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17783; J2A-MC-GZGD (Other: Eli Lilly and Company); QSC202755 (Other: Quotient Sciences); 2020-005750-15 (EudraCT Number)
Record Dates: First submitted 2021-09-16; First posted 2021-09-21 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04-15

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron; Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LY3502970 Prototype (Part A) (Experimental): Multiple doses of LY3502970 prototype administered orally.
  Interventions: Drug: LY3502970
- LY3502970 Reference (Part A) (Experimental): Multiple doses of LY3502970 reference administered orally.
  Interventions: Drug: LY3502970
- LY3502970 Prototype (Part B) (Experimental): Multiple doses of LY3502970 prototype administered orally.
  Interventions: Drug: LY3502970
- LY3502970 Reference (Part B) (Experimental): Multiple doses of LY3502970 reference administered orally.
  Interventions: Drug: LY3502970
- Esomeprazole (Part B) (Active Comparator): Multiple doses of Esomeprazole (Proton Pump Inhibitor) administered orally.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: LY3502970 — Administered orally.
  Arms: LY3502970 Prototype (Part A); LY3502970 Prototype (Part B); LY3502970 Reference (Part A); LY3502970 Reference (Part B)
Drug: Esomeprazole — Administered orally.
  Arms: Esomeprazole (Part B)

SUMMARY:
The main purpose of this study is to assess how fast LY3502970 gets into the blood stream and how long it takes the body to remove it when administered in multiple oral doses as new formulation compared to that of reference LY3502970 formulation. Information about safety and tolerability will be collected. The study is open to healthy participants. The study is conducted in two parts and it will last up to about 6 months, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation.
* Body mass index (BMI) of 18.5 to 35 kilograms per meter squared (kg/m²).

Exclusion Criteria:

* Have an abnormal blood pressure and/or pulse rate as determined by the investigator -minor deviations acceptable to investigator are allowed
* Have known liver disease, obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or have elevations in aminotransferases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) greater than 2X ULN (Upper Limit of Normal)
* Have an abnormality in the 12-lead ECG at screening that, in the opinion of the investigator, increases the risks associated with participating in the study
* Are women of child-bearing potential
* Are women who are lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3502970 | Predose up to 24 hours postdose
  PK: Cmax of LY3502970
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3502970 | Predose up to 24 hours postdose
  PK: AUC of LY3502970
PK: Time of Maximum Observed Concentration (Tmax) of LY3502970 | Predose up to 24 hours postdose
  PK: Tmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No